CLINICAL TRIAL: NCT05719662
Title: Effects of Weight Bearing Exercises With and Without Jaffrey's Core Stability Exercise Training on Dynamic Balance and Trunk Muscles Strength in Children With Down Syndrome.
Brief Title: Weight Bearing Exercises With and Without Jaffrey's Core Stability Exercise Training in Children With Down Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0748
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight bearing exercises (Experimental): weight bearing exercises (I.e standing on preferred foot, standing with close eyes, walking forward on a line using normal stride and heel to toe gait, stepping over response speed stick on balance beam).
  Interventions: Other: Weight bearing exercises
- Jaffrey's core stability exercises (Experimental): Jaffrey's core stability exercises (I.e contracting muscles, sitting on Swiss ball, Bridging, Squatting side lying bridge etc).
  Interventions: Other: Jaffrey's core stability exercises

INTERVENTIONS:
Other: Weight bearing exercises — Weight bearing exercises
  Arms: Weight bearing exercises
Other: Jaffrey's core stability exercises — Jaffrey's core stability exercises
  Arms: Jaffrey's core stability exercises

SUMMARY:
Down syndrome also known as trisomy 21, is a genetic disorder caused by the presence of all or part of a third copy of chromosome 21. It is usually associated with physical growth delays, mild to moderate intellectual disability, and characteristic facial features. There is no cure for Down syndrome. Education and proper care have been shown to improve quality of life. Some children with Down syndrome are educated in typical school classes, while others require more specialized education. Those with Down syndrome nearly always have physical and intellectual disabilities. They also typically have poor immune function and generally reach developmental milestones at a later age. They have an increased risk of a number of other health problems, including congenital heart defect, epilepsy, leukemia, thyroid diseases, and mental disorders. This study will determine effects of weight bearing exercises with and without Jaffery's core stability exercise training on dynamic balance and trunk muscles strength in children with Down syndrome. Randomized controlled study will be conducted in which data will be collected from children with down syndrome with calculated sample size of 18 which will randomly assigned into group A and group B. Group A would receive weight bearing exercises (I.e.

standing on preferred foot, standing with close eyes, walking forward on a line using normal stride and heel to toe gait, stepping over response speed stick on balance beam ).Group B would receive weight bearing exercises along with the jaffrey's core stability exercises (I.e.

contracting muscles, sitting on Swiss ball, Bridging, Squatting side lying bridge etc.).Frequency will be 5 sessions per week, of 1 hour and duration is of 5 months. Balance and trunk muscle strength will be pre assessed using pediatric balance scale and trunk control measurement scale respectively. The improvement will be measured with same tools. Data will be analyzed through SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Children with medical diagnosis of DS
* Age ranging from 4 to 10 year
* Both male and female genders
* Children who was able to stand and walk.

Exclusion Criteria:

* Any orthopedic limitation to exercise such as hip, knee, foot or spinal deformity.
* Children with planned orthopedic surgery in 6 months.
* Children with significantly impaired cognition.
* Children with hearing impairment

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric baalnce scale | 4 weeks
  Pediatric balance scale (PBS), is defined as the ability of a child to attain and maintain upright control. The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Trunk Control Measurement Scale | 4 weeks
  Trunk Control Measurement Scale is a clinical tool to measure trunk control in children

CONTACTS AND LOCATIONS:
Overall Officials: Sara Khan, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No